CLINICAL TRIAL: NCT06370793
Title: Ningbo Schizophrenia Cohort, a Longitudinal Population-based Ambispective Cohort Study
Brief Title: Ningbo Schizophrenia Cohort
Acronym: NSC
Status: Active, not recruiting | Type: Observational
Sponsor: Ningbo University (Other)
Collaborators: The Affiliated Kangning Hospital of Ningbo University (Unknown)
Responsible Party: Principal Investigator, Liya Liu, Associate Professor, Ningbo University
Other Study IDs: NBU-2024-011
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: Population-based healthcare database; Longitudinal study; Ambispective Cohort; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Schizophrenia
  Interventions: Other: Patient with schizophrenia without intervention

INTERVENTIONS:
Other: Patient with schizophrenia without intervention — Patients with schizophrenia identified based on exposures of interest to the study

SUMMARY:
In recent years, the prevalence of schizophrenia in China has continued to grow, and the burden of disease in society has continued to rise. In order to improve the prognosis of patients with schizophrenia and reduce the risk of disease relapse or readmission, researchers established a cohort based on the Ningbo Mental Health Information System in Ningbo, a sub-provincial city in the southern wing of the Yangtze River Delta of China, with a resident population of more than 9 million, and linked it to the residents' health records, and through the data linkage obtained data on patients in the full cycle of pre-onset, diagnosis, follow-up, disease changes and death, realising full-cycle management of patients with schizophrenia.

Currently, NSC has accumulated data on more than 30,000 patients with schizophrenia and obtained multi-dimensional longitudinal information through long-term follow-up and data linkage. All diseases follow the World Health Organization International Classification of Diseases 10th Edition (ICD-10) for clinical coding, and available data include baseline demographics, past history, family history, social functioning deficit screening scale scores, risk assessment, and so on and longitudinal health information from electronic health records (EHR), providing a solid data base for future real-world studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia (F20)
* Aged 18-65 years at the time of diagnosis

Exclusion Criteria:

* None.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were eligible if they were aged 18-65 years at diagnosis and had a diagnosis of schizophrenia confirmed by at least two independent visit records in the EHR. Additionally, they were required to provide signed informed consent, either personally or through their legal representatives, and possess complete electronic health records, including date of birth, gender, and a valid medical identifier. Subjects meeting any of the following criteria were not eligible to participate: (1) history of severe neurological diseases, including epilepsy, encephalitis, or brain tumours or (2) history of severe head trauma resulting in unconsciousness, to exclude trauma-induced psychotic symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 26899 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of circulatory system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records : Primary hypertension (I10), Cerebral infarction (I63), Transient cerebral ischaemic attacks and related syndromes (G45), Intracerebral haemorrhage (I61), Subarachnoid haemorrhage (I60), Hemorrhagic stroke (I60-I61), Stroke (I60-I64, I69), Pulmonary embolism (I26), Aortic aneurysm and dissection (I71), Cardiovascular disease (I20-I25), Atrial fibrillation (I48), Cardiomyopathy (I42), Peripheral vascular diseases (I73), Myocardial infarction (I21-I22), Heart failure (I50).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of endocrine system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records : Diabetes mellitus (E10-E14), Thyroid disorder (E00-E05, E61-E69, E07), Gout (E79, M10).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of pulmonary system and allergy diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records : Chronic pulmonary disease (J40-J47), Allergy (J30.1-J30.4, L23, L50.0, T78.0, T78.2, T78.4).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of gastrointestinal system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records : Ulcer/chronic gastritis (K22.1, K25-K28, K29.3-K29.5), Chronic liver disease (B16-B19, K70, K74, K76.6, I85), Inflammatory bowel disease (K50-K51), Diverticular disease of intestine (K57).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of musculoskeletal system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records :Connective tissue disorders (M05-M06, M08-M09, M30-M36, D86), Osteoporosis (M80-M82).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of urogenital system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records : Chronic kidney disease (N03, N11, N18-N19), Prostate disorders (N40).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of hematological system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records : HIV/AIDS (B20-B24), Anemias (D50-D53, D55-D59, D60-D61, D63-D64).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of cancers | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  Diagnosed with cancer (C00-C43, C45-C97) in electronic health records. Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of neurological system diseases | At least 1 year after being diagnosed with schizophrenia during the study period (2019-2023)
  At least one of the following diagnoses in the electronic health records :Vision problem (H40, H25, H54), Hearing problem (H90-H91, H93.1), Migraine (G43), Epilepsy (G40-G41), Parkinson's disease (G20-G22), Multiple sclerosis (G35), Neuropathies (G50-G64).
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of suicide | Recorded during the study period (2019-2023)
  At least one of the following records in the Ningbo Mental Health Information System: attempted suicide, suicide, death by suicide.
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.
Risk of violence | Recorded during the study period (2019-2023)
  At least one of the following records in the Ningbo Mental Health Information System: causing trouble, causing an accident, committing an offence, injuring another person.
  Calculation of Hazard ratios(HRs) with 95% confidence intervals, comparing the risk of illness in persons with schizophrenia with those without schizophrenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo University, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Ye H, Zhao Y, Li L, Qian Y, Zhu H, Bian G, Liu L. Ningbo Schizophrenia Cohort (NSC)-a longitudinal ambispective cohort based on electronic health records: cohort profile. BMJ Open. 2025 May 15;15(5):e091188. doi: 10.1136/bmjopen-2024-091188. PMID 40379328